#### The GlaxoSmithKline group of companies

| Division | ŀ | Worldwide Development |
|---|---|---|
| <b>Information Type</b> | | Clinical Pharmacology Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and analysis plan for a single dose study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of GSK1550188 in Chinese subjects with Systemic Lupus Erythematosus (SLE) |
|---|---|---|
| Compound Number | : | GSK1550188 |
| <b>Effective Date</b> | : | 02-MAY-2017 |

#### **Description:**

- The purpose of this reporting and analysis plan (RAP) is to describe the planned analyses and output to be included in the Clinical Pharmacology Study Report for Protocol 200909.
- This RAP is intended to describe some of the pharmacokinetic-pharmacodynamic analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the final Statistical Analysis Complete (SAC) deliverable.

**Subject:** Belimumab, intravenous, Systemic Lupus Erythematosus, Pharmacokinetics, Pharmacodynamics, Chinese subject.

#### **Author's Name and Functional Area:**

| PPD | | 28-APR-2017 |
|-------------|---------------|--------------|
| Statistics, | China Medical | (eSignature) |

#### Approved by:

| PPD | | 02-MAY-2017 |
|---------------|---------------|--------------|
| Statistics, C | China Medical | (eSignature) |

Copyright 2017 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **TABLE OF CONTENTS**

| 1. | INTRO | DUCTION | N | 4 |
|---|---|---|---|---|
| 2. | REPO | RTING & | ANALYSIS PLAN SYNPOSIS | 4 |
| 3. | SUMM<br>3.1.<br>3.2.<br>3.3.<br>3.4. | Changes<br>Study Ok<br>Study De | KEY PROTOCOL INFORMATIONs to the Protocol Defined Statistical Analysis Plan | 6<br>6<br>7 |
| 4. | PLANN<br>4.1.<br>4.2. | Interim A | LYSESalysesalyses | <mark>7</mark> |
| 5. | ANALY<br>5.1. | | PULATIONS Deviations | |
| 6. | | | SIDERATIONS FOR DATA ANALYSES AND HANDLING | 8 |
| 7. | STUD<br>7.1. | | ATION ANALYSESv of Planned Analyses | |
| 8. | PRIM <i>A</i><br>8.1. | | TISTICAL ANALYSES cokinetic Analyses Overview of Planned Pharmacokinetic Analyses Drug Concentration Measures Pharmacokinetic Parameters Statistical Analyses | 10<br>10<br>10 |
| 9. | SECO<br>9.1.<br>9.2. | Safety And 9.1.1. 9.1.2. Pharmac | TATISTICAL ANALYSES | 12<br>12<br>12<br>14 |
| 10. | REFE | RENCES. | | 15 |
| 11. | APPEN<br>11.1.<br>11.2.<br>11.3. | Appendix<br>11.1.1.<br>Appendix<br>11.2.1.<br>11.2.2. | C 1: Time & Events | 1720202121 |

#### **CONFIDENTIAL**

| | | 11.3.2.2. | Derivations and Handling of Missing Baseline | |
|---|---|---|---|---|
| | | | Data | 21 |
| | 11.3.3. | Reporting | Process & Standards | <mark>22</mark> |
| 11.4. | Appendi | x 4: Derive | d and Transformed Data | 2 <mark>5</mark> |
| | 11.4.1. | | | |
| | 11.4.2. | Study Pop | oulation | 2 <mark>5</mark> |
| | 11.4.3. | | | |
| | 11.4.4. | | okinetic | |
| | 11.4.5. | Pharmaco | odynamic or Biomarker | 26 |
| | 11.4.6. | | okinetic/Pharmacodynamic | |
| 11.5. | Appendi | x 5: Prema | ture Withdrawals & Handling of Missing Data | 28 |
| | 11.5.1. | Premature | e Withdrawals | 28 |
| | 11.5.2. | | of Missing Data | |
| | | | Handling of Missing Dates | |
| | | | Handling of Partial Dates | |
| 11.6. | | | Laboratory Evaluations | |
| 11.7. | | | viations & Trade Marks | |
| | 11.7.1. | | ions | |
| | | | ks | |
| 11.8. | Appendi | | Data Displays | |
| | 11.8.1. | | lay Numbering | |
| | 11.8.2. | | mple Referencing | |
| | 11.8.3. | | le [Priority] | |
| | 11.8.4. | Study Pop | oulation Tables | 34 |
| | 11.8.5. | | bles | |
| | 11.8.6. | | okinetic Tables | |
| | 11.8.7. | Pharmaco | odynamic Tables | 39 |
| | 11.8.8. | | jures | |
| | 11.8.9. | Pharmaco | okinetic Figures | 40 |
| | 11.8.10. | | odynamic Figures | |
| | | | gs | |
| | | | Listings | |
| 11.9. | Appendi | x 9: Examp | le Mock Shells for Data Displays | 46 |

### 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Pharmacology Study Report for Protocol:

All decisions regarding key analysis, as defined in this RAP document, have been made prior to first subject first visit (FSFV).

# 2. REPORTING & ANALYSIS PLAN SYNPOSIS

| Overview | Key Elements of the Reporting and Analysis Plan |
|---|---|
| Purpose | The purpose of this Reporting and Analysis Plan (RAP) is to describe: |
| | All planned analyses and outputs required for the final Clinical<br>Pharmacology Study Report (CPSR) of study 200909 |
| Protocol | This RAP is based on the protocol (Dated: 26/JAN/2016) of study 200909 (GSK Document Number 2013N175219_00). |
| Primary<br>Objective | To investigate the pharmacokinetics (PK) of intravenously (IV) administered GSK1550188 10 mg/kg in Chinese subjects with SLE. |
| Secondary<br>Objective | To evaluate the safety and tolerability of GSK1550188 in Chinese subjects with SLE. |
| | To investigate the effect of GSK1550188 on pharmacodynamics (PD) of B cell subsets. |
| Primary<br>Endpoint | • Serum concentrations and the derived pharmacokinetic parameters of GSK1550188: Cmax, t1/2, AUC(0-t), AUC(0-∞), λz , CL and Vz. |
| Secondary<br>Endpoint | Safety and tolerability endpoints: adverse events, vital sign, 12-lead ECG, and clinical laboratory safety tests |
| | B cell subsets (CD20+, CD20+/27+ memory, CD20+/27-naïve, CD20+/69+ activated, CD20+/138+ plasmacytoid, CD19+/27BRIGHT/38BRIGHT SLE subset and CD20-/138+ plasma cells) |
| Study<br>Design | Multicenter, single dose study of intravenous GSK1550188 at a dose of 10 mg/kg Chinese subjects with SLE. |
| | A medical screen within 30 days prior to the first dose. |
| | • Subjects will receive the dose on Day 0 and be kept in the study center up to 24 hours post dosing with subsequent outpatient visits occurring on Days 1, 7, 14, 21, 28, 42, 56, and 84. |
| Planned | No interim analyses are planned. |
| Analyses | The final planned analyses will be performed after all subjects have completed the study and after database freeze (both the CRF data and PK data). |
| Analysis | The 'Safety' Population (Comprised of subjects who receive at least |

| Overview | Key Elements of the Reporting and Analysis Plan |
|---|---|
| Population | one dose of study medication) will be used to evaluate Study Population and Safety. |
| | • The 'Pharmacokinetic Concentration Population' (Comprised of subjects who receive the study medication and for whom a pharmacokinetic sample is obtained and analysed). |
| | • The 'Pharmacokinetic Parameter Population' is defined as all subjects who receive a dose of GSK1550188 and for whom pharmacokinetic parameters can be calculated. |
| | • The 'Pharmacodynamic Population' is defined as all subjects who receive the study medication and for whom pharmacodynamic data is available. |
| Hypothesis | There is no formal hypothesis being tested in this study. |
| Primary<br>Analyses | • Pharmacokinetics: Pharmacokinetic data will be presented in graphical and/or tabular form and will be summarized descriptively. |
| Secondary<br>Analyses | Safety data will be presented in tabular and/or graphical format and summarized descriptively according to GSK's Integrated Data Standards Library (IDSL) standards. |
| | Pharmacodynamics data of B cell subsets will be listed and summarized. |
| | • Other exploratory PK-PD analyses will be considered, when appropriate. These include exposure (PK parameters and concentrations)-response (B-cell subsets) analyses using linear and nonlinear mixed effect modelling methods. The results may be summarized in a report, separate from the main CPSR. |

# 3. SUMMARY OF KEY PROTOCOL INFORMATION

# 3.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol (Dated: 26/JAN/2016).

# 3.2. Study Objective(s) and Endpoint(s)

| Ob | jectives | Endpoints |
|---|---|---|
| Pri | mary | Primary |
| • | To investigate the pharmacokinetics (PK) of intravenously (IV) administered GSK1550188 10 mg/kg in Chinese subjects with SLE | • Serum concentrations and the derived pharmacokinetic parameters of GSK1550188: Cmax, t1/2, AUC(0-t), AUC(0-∞), λz, CL and Vz. |
| Sec | condary Objectives | Secondary Endpoints |
| • | To evaluate the safety and tolerability of GSK1550188 in Chinese subjects with SLE. | • Safety and tolerability endpoints: adverse events, vital sign, 12-lead ECG, and clinical laboratory safety tests. |
| • | To investigate the effect of GSK1550188 on the pharmacodynamics (PD) of B cell subsets. | B cell subsets (CD20+, CD20+/27+<br>memory, CD20+/27-naïve, CD20+/69+<br>activated, CD20+/138+ plasmacytoid,<br>CD19+/27BRIGHT/38BRIGHT SLE<br>subset and CD20-/138+ plasma cells). |

### 3.3. Study Design



# 3.4. Statistical Hypotheses

No formal hypothesis is being tested in the study.

#### 4. PLANNED ANALYSES

### 4.1. Interim Analyses

No interim analyses are planned.

# 4.2. Final Analyses

The final planned analyses will be performed after all subjects have completed the study and after database freeze (both the CRF data and PK data).

#### 5. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Safety | Subjects who receive at least one dose | Study Population |
| | of study medication. | • Safety |
| Pharmacokinetic | Subjects who receive the study | PK Analyses |
| Concentration | medication and for whom a | |
| Population | pharmacokinetic sample is obtained | |
| | and analysed. | |
| Pharmacokinetic | Subjects who receive a dose of | PK Analyses |
| Parameter | GSK1550188 and for whom | |
| Population | pharmacokinetic parameters can be | |
| | calculated. | |
| Pharmacodynamic | Subjects who receive the study | PD Analyses |
| Population | medication and for whom | |
| | pharmacodynamic data are available. | |

#### 5.1. Protocol Deviations

- A listing of the inclusion/exclusion criteria deviation record for all subjects with deviations will be provided.
- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarized and listed.
- Other deviations will be noted as applicable, including use of prohibited concomitant medications during the study, incorrect study drug administration, and any other deviations deemed to have the potential for notably influencing the study results.
- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
  - o This dataset will be the basis for listing of protocol deviations.

For details of important protocol deviations criteria please refer to protocol deviation management plan.

# 6. GENERAL CONSIDERATIONS FOR DATA ANALYSES AND HANDLING CONVENTIONS

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|---|---|
| Section 11.1 | Appendix 1: Time & Events |
| Section 11.2 | Appendix 2: Treatment States |
| Section 11.3 | Appendix 3: Data Display Standards & Handling Conventions |
| Section 11.4 | ection 11.4 Appendix 4: Derived and Transformed Data |
| Section 11.5 | Appendix 5: Premature Withdrawals & Handling of Missing Data |
| Section 11.6 | Appendix 6: Clinical Laboratory Evaluations |

#### 7. STUDY POPULATION ANALYSES

# 7.1. Overview of Planned Analyses

The Safety Analyses will be based on the Safety population, unless otherwise specified. Screen failures will be listed and summarized for all 'Screened' subjects.

The Pharmacokinetic Analyses will be based on the Pharmacokinetic concentration population and Pharmacokinetic parameter population.

The Pharmacodynamic Analyses will be based on the Pharmacodynamic population.

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 8 (Section 11.8): List of Data Displays.

Table 2 Overview of Planned Study Population Analyses

| Display Type | Data | Data Display's Generated | |
|---|---|---|---|
| | Figure | Table | Listing |
| Subject Disposition | | | |
| Subject Disposition | | Υ | |
| Reasons for Screening Failures | | Υ | Y |
| Reasons for Withdrawals | | | Y |
| Study Analysis Populations | | Υ | Y |
| Inclusion and Exclusion Criteria Deviations | | | Y |
| Important Protocol Deviations | | Υ | Y |
| Other Protocol Deviations | | Υ | Υ |
| Demography | • | | |
| Demographics Characteristics | | Υ | Y |
| Race and Racial Combinations | | | Υ |

| Display Type | Data Display's Generated | | |
|---|---|---|---|
| | Figure | Listing | |
| Medical Condition & Concomitant Medications | | | |
| Concomitant Medication | | | Υ |
| Medical Conditions (Current/Past) | | | Υ |

#### NOTES:

• Y = Yes display generated.

#### 8. PRIMARY STATISTICAL ANALYSES

### 8.1. Pharmacokinetic Analyses

### 8.1.1. Overview of Planned Pharmacokinetic Analyses

The pharmacokinetic (PK) concentration and parameter analyses will be based on the PK concentration and parameter population, unless otherwise specified.

Table 3 provides an overview of the planned analyses, with full details being presented in Appendix 8: List of Data Displays.

Table 3 Overview of Planned Pharmacokinetic Analyses

| [Endpoint / | | Untrans | sformed | | Log-Transformed | | | |
|---|---|---|---|---|---|---|---|---|
| Parameter/ Display | Sumr | mary | Indiv | <i>r</i> idual | Sum | nmary | Individual | |
| Type] | T F | | F | L | T | F | F | L |
| PK Concentration Data | | | | | | | | |
| Plasma Drug | V | V | V | V | | V | V | |
| Concentrations | ī | Ī | Ĭ | Ĭ | | Ĭ | T | |
| PK Parameter Data | | | | | | | | |
| Parameters | Υ | | | Υ | Υ | | | Υ |

#### NOTES:

- T = Table, F = Figure, L = Listings, Y = Display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 8.1.2. Drug Concentration Measures

Refer to Appendix 3: Data Display Standards & Handling Conventions (Section 11.3.3 Reporting Process & Standards).

#### 8.1.3. Pharmacokinetic Parameters

• Refer to Appendix 3: Data Display Standards & Handling Conventions (Section 11.3.3 Reporting Process & Standards).

- The pharmacokinetic parameters will be calculated by standard noncompartmental analysis according to current working practices and usingWinNonlin6.3 or above.
- All calculations of non-compartmental parameters will be based on actual sampling times.
- If data permits, population PK modelling will be conducted and independent PK modelling plan document may be provided.
- Pharmacokinetic parameters described as following and in Table 4 will be determined from intravenously (IV) administered GSK1550188, as data permits.

| Table 4 | Derived | Pharmaco | kinetic | <b>Parameters</b> |
|---------|---------|----------|---------|-------------------|
|---------|---------|----------|---------|-------------------|

| Parameter | Parameter Description |
|---|---|
| AUC(0−∞) | Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time |
| AUC(0-t) | Area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration |
| CL | Clearance |
| Cmax | Maximum observed concentration |
| λz | Terminal phase rate constant |
| $t_{1/2}$ | Terminal phase half-life |
| Vz | Volume of distribution after intravenous administration |

#### 8.1.4. Statistical Analyses

Pharmacokinetic concentration and parameter data will be summarized descriptively and presented in tabular and/or graphic formats per GSK IDSL standard.

All derived pharmacokinetic parameters described above will be summarised and listed according to the Pharmacokinetic Parameter Population defined in Section 5. For each of these parameters the following summary statistics will be calculated: arithmetic mean, 95% confidence interval for the arithmetic mean, standard deviation, median, minimum, maximum, between coefficient of variation, geometric mean, 95% confidence interval for the geometric mean and standard deviation of log-transformed data.

For the purposes of calculating summary statistics and for statistical analysis, all PK parameters will be log-transformed.

Between subjects coefficient of variation (%CVb) for log-transformed data will be calculated according to the following methods:

$$\%CVb = SQRT(exp(SD^2)-1) * 100$$

where SD is the standard deviation of the log-transformed data.

Between subjects coefficient of variation (%CVb) for untransformed data will be calculated according to the following methods:

%CVb = (SD/Mean) \* 100

#### 9. SECONDARY STATISTICAL ANALYSES

#### 9.1. Safety Analyses

#### 9.1.1. Overview of Adverse Events

The CRF texts for adverse events (AEs) will be coded using MedDRA version 19.0 or above, and will be reported using the System Organ Class (SOC) and Preferred Term (PT). In the summary of AEs, the incidence of AEs will be the number of subjects reporting AEs and not the number of AEs reported. Multiple occurrences of the same AE in one individual will be counted only once when calculating the number and percentage of subjects.

The following AEs will be summarized and listed:

- All AEs;
- All AEs by maximum intensity
- All drug-related AEs
- All drug-related AEs by maximum intensity
- All Serious AEs
- All AEs leading to study withdrawals

More details can be found in Section 9.1.2.

#### 9.1.2. Overview of Planned Safety Analyses

The safety analyses will be based on the "Safety population", unless otherwise specified. Table 5 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 8: List of Data Displays.

Table 5 Overview of Planned Safety Analyses

| [Endpoint / Parameter/ | | Abs | olute | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|
| Display Type] | Sum | ımary | | /idual | | mary | Indiv | vidual |
| | Т | F | F | L | Т | F | F | L |
| Exposure | | | | | | | | |
| Exposure | | | | Υ | | | | |
| Adverse Events | | | | | | | | |
| All AEs [1] | Υ | | | Υ | | | | |
| AEs – Max Intensity | Υ | | | Υ | | | | |
| Drug Related AEs | Υ | | | Υ | | | | |
| Drug Related AEs – Max | Y | | | Y | | | | |
| Intensity | | | | | | | | |
| Serious AEs | | | | Υ | | | | |
| AEs leading to study | | | | Υ | | | | |
| Withdrawal | | | | | | | | |
| Laboratory Values | T | | 1 | T | 1 | T | 1 | Т |
| Clinical Chemistry | Y | | | Υ | Y | | | |
| Hematology | Υ | | | Υ | Y | | | |
| Urinalysis | Y | | | Y | | | | |
| Immunoglobulin | Υ | | | Υ | Y | | | |
| Toxicity Grade <sup>[2]</sup> : | Υ | | | | Y | | | |
| Chemistry | | | | | | | | |
| Toxicity Grade: | Y | | | | Υ | | | |
| Hematology | ., | | | | | | | |
| Toxicity Grade: Urinalysis | Y | | | | Y | | | |
| Toxicity Grade: | Y | | | | Y | | | |
| Immunoglobulin | | | L | | | | | |
| ECC Peremeters | Υ | | I | | I | I | | T |
| ECG Parameters | Ť | | | V | Υ | | | |
| ECG Values | V | | | Y | Y | | | |
| Abnormal ECG | Y | | | Υ | | | | <u> </u> |
| Vital Signs | | | | | \ \\ \ | | | |
| Vital Values | Υ | | <u> </u> | Υ | Y | | | <u> </u> |
| Liver Events | | | | | | 1 | 1 | |
| Liver Events | | | | Υ | | | ] | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated, PCI=Potential Clinical Importance
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. Listing will include subject's numbers for individual AE's & the table includes AE system organ classes and preferred terms.
- 2. Toxicity grades are defined in Appendix 3 of the protocol.

### 9.2. Pharmacodynamic Analyses

### 9.2.1. Overview of Planned Pharmacodynamic Analyses

The pharmacodynamic analyses will be based on the "pharmacodynamic population", unless otherwise specified. Table 6 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 8: List of Data Displays.

Table 6 Overview of Planned Pharmacodynamic Analyses

| [Endpoint / | | Absolute | | Change from Baseline | | |
|---|---|---|---|---|---|---|
| Parameter/ Display<br>Type] | Figure | Table | Listing | Figure | Table | Listing |
| B Cell Subsets | Υ | Υ | Υ | Υ | Υ | |

#### NOTES:

T = Table, F = Figure, L = Listings, Y = Display generated.

### 9.2.2. Pharmacokinetic-Pharmacodynamic Modelling Analyses

Supplemental compartmental PK modelling and additional PK/PD modelling analyses may be conducted to characterize the relationship between Belimumab exposure and the B cell subsets profile. These supplemental analyses, as feasible, will be outlined and reported in a separate document.

# 10. REFERENCES

Human Genome Sciences Clinical Pharmacokinetics Report HGS1006-POPPK. Population pharmacokinetics of belimumab (monoclonal anti-BLyS antibody) following intravenous administration in patients with systemic lupus erythematosus. March, 2010.

# 11. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 6 | : General Considerations for Data Analyses & Data Handling Conventions |
| Section 11.1 | Appendix 1: Time and Events |
| Section 11.2 | Appendix 2: Treatment States |
| Section 11.3 | Appendix 3: Data Display Standards & Handling Conventions |
| | Study Treatment & Sub-group Display Descriptors |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 11.4 | Appendix 4: Derived and Transformed Data |
| | General, Study Population & Safety |
| | Pharmacokinetic |
| | Pharmacodynamic or Biomarkers |
| | Pharmacokinectic/Pharmacodynamic |
| Section 11.5 | Appendix 5: Premature Withdrawals & Handling of Missing Data |
| | Premature Withdrawals |
| | Handling of Missing Data |
| Section 11.6 | Appendix 6: Clinical Laboratory Evaluations |
| Other RAP Appendices | |
| Section 11.7 | Appendix 7: Abbreviations & Trade Marks |
| Section 11.8 | Appendix 8: List of Data Displays |

# 11.1. Appendix 1: Time & Events

# 11.1.1. Protocol Defined Time & Events

| Visit | 1 | | | | 2 | | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day | Screening<br>Day -30 to -1 | Pre | 0 | Da<br>5m | ay 0<br>1h | 6h | 24h | Day<br>1 | Day<br>7 | Day<br>14 | Day<br>21 | Day<br>28 | Day<br>42 | Day<br>56 | Day<br>84 | Discontinuation <sup>9</sup> |
| Informed consent <sup>1</sup> | x | | | | | | | | | | | | | | | |
| Medical History | х | х | | | | | | | | | | | | | | |
| Demography | х | | | | | | | | | | | | | | | |
| Complete physical examination, including Height | х | | | | | | | | | | | | | | | |
| Inclusion/Exclusion criteria | х | | | | | | | | | | | | | | | |
| Body weight | | х | | | | | | | | | | | | | | |
| Vital signs <sup>2</sup> | х | х | | Х | Х | Х | х | х | Х | Х | Х | Х | Х | х | Х | х |
| Record Concomitant<br>Medications | Х | х | х | Х | Х | Х | х | х | х | Х | Х | х | Х | х | Х | х |
| Clinical Laboratory test <sup>3</sup> | Х | х | | | | | х | | | х | | х | | х | х | х |
| Spot urine (protein to | х | | | | | | | | | | | | | | | |

| Visit | 1 | | | | 2 | | | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day | Screening | | | | ay O | 1 | ı | Day | Day | Day | Day | Day | Day | Day | Day | Discontinuation <sup>9</sup> |
| | Day -30 to -1 | Pre | 0 | 5m | 1h | 6h | 24h | 1 | 7 | 14 | 21 | 28 | 42 | 56 | 84 | |
| creatinine ratio) | | | | | | | | | | | | | | | | |
| Urine drug/alcohol screen | Х | | | | | | | | | | | | | | | |
| HIV, Hepatitis B, C4 | Х | | | | | | | | | | | | | | | |
| Pregnancy test (women) <sup>5</sup> | х | х | | | | | | | | | | Х | | | Х | Х |
| Chest X ray | х | | | | | | | | | | | | | | | |
| 12 lead ECG | Х | х | | | | | х | | | | | | | | Х | х |
| Biological Markers <sup>6</sup> | X <sup>7</sup> | х | | | | | | | | Х | | Х | Х | Х | Х | |
| Blood PK sampling | | Х | | х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | |
| AE/SAE Review <sup>8</sup> | Х | Х | Х | х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | х |
| Admission to Unit | | Х | | | | | | | | | | | | | | |
| Dosing | | | х | | | | | | | | | | | | | |
| Discharge | | | | | | | Х | | | | | | | | | |
| Outpatient Visit | Х | | | | | | | Х | Х | Х | Х | Х | Х | Х | Х | х |

- 1. Each subject must sign an informed consent form prior to undergoing any Screening assessments.
- 2. Vital signs include temperature, sitting blood pressure and heart rate.
- 3. Clinical Laboratory test include hematology, chemistry and urinalysis (including CRP and Erythrocyte Sedimentation Rate on screening). ALT and/or AST elevations of greater than 2.5 x ULN will require additional Hepatitis B assessment, see Section 6.2.1.1 in protocol.
- 4. HIV antibody, Hepatitis B surface antigen, anti-HBc and Hepatitis C antibody.
- 5. Pregnancy should be assessed with a blood test at Screening and with a urine test during the treatment period.
- 6. Biomarkers include immunoglobulins B cell subsets (CD20+, CD20+/27+ memory, CD20+/27-naïve, CD20+/69+ activated, CD20+/138+ plasmacytoid, CD19+/27BRIGHT/38BRIGHT SLE subset and CD20-/138+ plasma cells).
- 7. Only immunoglobulins (IgG, IgM and IgA) and autoantibodies (anti-dsDNA, ANA).
- 8. Includes subject history to be reported on CRF regarding any general signs or symptoms of infection.
- 9. If a subject prematurely withdraws for any reason, the investigator must make every effort to assess the items specified on discontinuation test.

# 11.2. Appendix 2: Treatment States

Assessments and events will be classified according to time of occurrence relative to the start and/or stop date of the study treatment.

#### 11.2.1. Treatment States for Concomitant Medications Data

No definition of treatment states for concomitant medications in this study.

#### 11.2.2. Treatment States for AE Data

| Treatment State | Definition |
|---|---|
| Onset Time Since start time of dosing | AE Onset Date – Dosing Start Date + 1 |
| Duration (Days) | AE Resolution Date – AE Onset Date + 1 |
| Drug-related | If relationship is marked 'YES' on Inform/CRF OR value is missing. |

#### NOTES:

• If the study treatment stop date is missing then the AE will be considered to be On-Treatment.

# 11.3. Appendix 3: Data Display Standards & Handling Conventions

#### 11.3.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | |
|---|---|
| Description Data Displays for Reporting | |
| Belimumab 10 mg/kg | Belimumab 10 mg/kg |

#### 11.3.2. Baseline Definition & Derivations

#### 11.3.2.1. Baseline Definitions

For all endpoints (expect as noted in the table) the baseline value will be the last pre-dose assessment. The change from baseline will be calculated by subtracting the baseline values from the individual post-baseline values. If either the baseline or post-baseline value is missing, the change from baseline is set to missing as well.

Table 7 Baseline Definitions

| Devemeter | | Study Assessments Considered As Baseline | | |
|---|---|---|---|---|
| Parameter | Screening | Screening Day -1 | | Data Display |
| Safety | · | | | |
| LAB | Х | | Х | Day 0(Pre Dose)[1] |
| Vital Signs | Х | | Х | Day 0 (Pre Dose) |
| 12 Lead ECG | X | | Х | Day 0 (Pre Dose) |

#### NOTES:

- Unless otherwise stated, the mean of replicate assessments at any given time point will be used as the value for that time point.
- 1. For baseline value, if it is missing at baseline visit, then the latest non-missing value of screening will be used to replace.

#### 11.3.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|---|---|
| Change from Baseline | = Post-Dose Visit Value – Baseline |
| % Change from Baseline | = 100 x [(Post-Dose Visit Value – Baseline) / Baseline] |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 11.3.2.1. Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.
- The baseline definition will be footnoted on all change from baseline displays.

#### 11.3.3. Reporting Process & Standards

| Reporting Process | |
|---|---|
| Software | |
| The currently supported versions of SAS software will be used. | |
| Reporting Area | |
| HARP Server | US |
| HARP Area | : \ARPROD\GSK1550188\200909\Final |
| QC Spreadsheet | : \ARWORK\GSK1550188\200909\Final\Documents |
| Analysis Datasets | |

- Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.1.3 & AdaM IG Version 1.0).
- For creation of ADaM datasets (ADCM/ADAE), the same version of dictionary datasets will be implemented for conversion from SI to SDTM.

#### **Generation of RTF Files**

RTF files will be generated.

#### **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses :
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.

#### **Reporting Standards**

- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures, summaries and statistical analyses.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables.
- Unscheduled visits will not be included in figures.
- All unscheduled visits will be included in listings.

| | Descriptive Summary Statistics | |
|---|---|---|
| Continuous Data Refer to IDSL Statistical Principle 6.06.1 | | Refer to IDSL Statistical Principle 6.06.1 |
| | Categorical Data | N, n, frequency, % |

#### **Reporting of Pharmacokinetic Concentration Data**

| Descriptive | Summary |
|-------------|---------|
| Statistics | |

Refer to IDSL Statistical Principle 6.06.1

Refer to GUI\_51487

Any plasma concentrations below the assay lower limit of quantification (NQ) will be imputed using the following rules:

- NQs at the beginning of a subject profile (i.e. before the first incidence of a measurable concentration) are deemed to be zero as it is assumed that in this circumstance no drug is yet measurable in the plasma.
- For NQs at the end of the subject profile (i.e. after the last incidence of a measurable concentration):
  - (1) for individual plots and pharmacokinetic analyses these are dropped (set to missing) as they do not provide any useful information (and can erroneously indicate that absolutely no drug is present)
  - (2) for summary statistics these are set to 0 (to avoid skewing of the summary statistics)
- Individual NQs which fall between two measurable concentrations are set to missing (individual values of this nature are assumed to be an anomaly)
- More than one consecutive NQ between measurable concentrations are set to 0.
- Measurable concentrations after more than one consecutive midprofile NQ (a mid-profile NQ is defined as any NQ where measurable concentrations exist both before and after that NQ in the profile):

For summary, these will be set to missing.

For individual plot, no action will be done.

All NQs will remain as "NQ" in listings.

| Reporting Standards | |
|---|---|
| Reporting of Pharmacokinetic Parameters | |
| Descriptive Summary<br>Statistics.<br>(Log Transformed) | N, n, arithmetic mean, median, min, max, SD, 95% CI of arithmetic mean will be provided for non-logged data. For logged data, N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) of logged data and between geometric coefficient of variation (CVb (%)) will be reported. [1] CVb (%) = √ (exp(SD²) - 1) * 100 [NOTE: SD = SD of log transformed data] |
| Reporting of Pharmacodynamic Data | |
| Descriptive Summary<br>Statistics. (Not Being<br>Log Transformed) | B cell subsets (CD20+, CD20+/27+ memory, CD20+/27-naïve, CD20+/69+ activated, CD20+/138+ plasmacytoid, CD19+/27BRIGHT/38BRIGHT SLE subset and CD20-/138+ plasma cells) |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

### 11.4. Appendix 4: Derived and Transformed Data

#### 11.4.1. General

#### **Multiple Measurements at One Time Point**

- Where multiple measurements are recorded for a particular time point, the mean of the measurements will be calculated and used in any derivation of summary statistics. However all available data will be listed.
- Where more than the specified number of measurements has been taken, the recorded values nearest to the scheduled time will be used in the derivation of the appropriate summary measure (i.e. mean or maximum).

#### **Study Day**

- The Study day will be provided on the listings to show the relative date to a reference date. In this study, the reference date will be defined as the date of visit on Day 0 (i.e. start date of dosing). The study day will be calculated by:
  - Date of interest ≥ Date of visit on Day 0
     Study Day = Date of interest –Date of visit on Day 0+1
  - Date of interest < Date of visit on Day 0</li>
     Study Day = Date of interest –Date of visit on Day 0

### 11.4.2. Study Population

#### **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any subject with a missing day will have this imputed as day '15'.
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.
- Use informed consent date as Reference for age calculation.

#### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)]<sup>2</sup>

### 11.4.3. Safety

#### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Significant Digits = '< x ' becomes x 0.01
  - Example 2: 1 Significant Digit = '> x' becomes x + 0.1
  - Example 3: 0 Significant Digits = '< x' becomes x 1

#### 11.4.4. Pharmacokinetic

#### PK

Descriptive statistics (N, mean, SD, median, minimum, and maximum) will be used to summarize the concentration values of belimumab in plasma at each sampling time point / collection interval for each profile day. Individual subject concentration data will be listed.

Individual plasma concentration-time profiles and median/mean profiles will be plotted. Each of the figures will contain one plot on the untransformed scale (i.e. a linear plot) and one plot on the log transformed scale (i.e. log-linear plot).

The concentration data described above will be summarised, listed and plotted based on Pharmacokinetic Concentration Population defined in Section 5.

The pharmacokinetic parameters (AUC(0- $\infty$ ), AUC(0-t), C<sub>max</sub>, t<sub>½</sub>,  $\lambda$ z, CL, Vz) will be determined from the plasmaconcentration-time data for belimumab. The pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using WinNonlin6.3 or above. All calculations of non-compartmental parameters will be based on actual sampling times.

All the derived parameters described above will be summarised and listed. For each of these parameters the following summary statistics will be calculated: arithmetic mean, 95% confidence interval for the arithmetic mean, standard deviation, median, minimum, maximum, between coefficient of variation, geometric mean, 95% confidence interval for the geometric mean and standard deviation of log-transformed data.

All derived pharmacokinetic parameters described above will be summarised and listed according to the Pharmacokinetic Parameter Population defined in Section 5.

### 11.4.5. Pharmacodynamic or Biomarker

#### PD

The central laboratory will transmit the following results electronically to GlaxoSmithKline:

 B cell subsets (CD20+, CD20+/27+ memory, CD20+/27- naïve, CD20+/69+activated, CD20+/138+ plasmacytoid, CD19+/27BRIGHT/38BRIGHT SLE subset and CD20-/138+ plasma cells).

Estimates of percent change from baseline for B cell subsets will be performed in the PD population. The 6-point summary, n, mean, median, standard deviation, minimum and maximum will be used for analysis. All derived parameters will be listed and summarized.

The mean and median profile of raw data of B cell subsets will be figured using line plots by treatment. The plots with the level of B cell subsets on y-axis and the planned time on x-axis will be prepared.

# 11.4.6. Pharmacokinetic/Pharmacodynamic

### PK/PD

Other exploratory PK-PD analyses will be considered, when appropriate. These include exposure (PK parameters and concentrations)-response (B-cell subsets) analyses using linear and nonlinear mixed effect modelling methods. The results may be summarized in a report, separate from the main CPSR.

# 11.5. Appendix 5: Premature Withdrawals & Handling of Missing Data

# 11.5.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as completion of all the phases of the study including the follow up visit.</li> <li>Withdrawn subjects were not replaced in the study.</li> <li>All subjects who withdraw prematurely from the study will be documented and the reason for their withdrawal recorded in the final Clinical Pharmacology Study</li> </ul> |
| | <ul> <li>Report (CPSR).</li> <li>All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary, tables and figures, unless otherwise specified.</li> </ul> |
| | <ul> <li>In the event that the study is prematurely discontinued, all available data will be<br/>listed and a review carried out by the study team to assess which statistical<br/>analyses are still considered appropriate and population approach may be used<br/>to deal with such situations as appropriate.</li> </ul> |

# 11.5.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> </ul> </li> </ul> |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 11.5.2.1. Handling of Missing Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing. |

# 11.5.2.2. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Concomitant<br>Medications | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year).</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |
| Adverse<br>Events | <ul> <li>Any partial dates for adverse events will be raised to data management. If the full date cannot be ascertained, the following assumptions will be made: <ul> <li>If the partial date is a start date, a '01' will be used for the day.</li> <li>However, if these results in a date prior to start date of study treatment and the event could possibly have occurred on treatment from the partial information, then the start date of study treatment will be assumed to be the start date.</li> <li>The AE will then be considered to start on-treatment (worst case).</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year).</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 11.6. Appendix 6: Clinical Laboratory Evaluations

#### **Character Values**

For laboratory values that are above or below the lower limit of quantification, having only character values starting with "<" or ">," numeric values will be derived using the following rules, where LRESSI is the character result in standard units, and LNRES is the numeric version of the result:

- If LRESSI > x then LNRES = x + 1, where x is an integer >= 1.
   If LRESSI > x.y then LNRES = x.y +0.1, where x, y are integers.
   If LRESSI > x.yz then LNRES = x.yz + 0.01, where x, y, z are integers.
   Etc.
- If LRESSI "< x" then LNRES = x 1, where x is an integer >= 1.
   If LRESSI "< x.y" then LNRES = x.y 0.1, where x, y are integers.</li>
   If LRESSI "< x.yz" then LNRES = x.yz 0.01, where x, y, z are integers.</li>
   Etc.

#### **Severity Grade**

The laboratory value severity grade tables are showed in Appendix 3 of protocol. Laboratory toxicity will be graded using Adverse Event Severity Grading Tables when possible. Note that four analytes, potassium, glucose, calcium, and sodium, have toxicities in both the high and low directions, and both will be presented in toxicity displays by the name of the toxicity. For example, calcium will have two toxicity sections, one for hypocalcaemia and one for hypercalcaemia. These toxicities will be mapped to their high or low form by using the following formulae:

RESULT 
$$<$$
 (LLN+ULN)/2 = "Hypo" toxicity

RESULT 
$$> (LLN+ULN)/2 = "Hyper" toxicity$$

where LLN is Lower Limit of Normal and ULN is Upper Limit of Normal.

# 11.7. Appendix 7: Abbreviations & Trade Marks

# 11.7.1. Abbreviations

| AE | Adverse event |
|---|---|
| ALT | Alanine aminotransferase |
| AST | Aspartate aminotransferase |
| AUC | Area under concentration-time curve |
| AUC(0-∞) | Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time |
| AUC(0-t) | Area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration |
| BMI | Body mass index |
| BP | Blood pressure |
| CL | Clearance |
| Cmax | Maximum observed concentration |
| CRF | Case report form |
| %CV | Coefficient of variation |
| ECG | Electrocardiogram |
| GSK | GlaxoSmithKline |
| HBsAg | Hepatitis B surface antigen |
| hr | hour |
| IV | Intravenous |
| kg | Kilogram |
| mg | Milligram |
| mL | Millilitre |
| msec | Millisecond |
| ng | Nanogram |
| PK | Pharmacokinetics |
| RBC | Red blood cell |
| SAE | Serious adverse event(s) |
| SD | Standard deviation |
| λz | Terminal phase rate constant |
| t1/2 | Terminal phase half-life |
| ULN | Upper limit of normal |
| WBC | White blood cell |
| Vz | Volume of distribution after intravenous administration |
| | Volume of distribution after intravenous administration at steady state |

### 11.7.2. Trademarks

Trademarks of the GlaxoSmithKline Group of Companies

BELIMUMAB

Trademarks not owned by the GlaxoSmithKline Group of Companies

SAS

WinNonlin

# 11.8. Appendix 8: List of Data Displays

#### 11.8.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|--------------|------------|
| Study Population | 1.01 to 1.07 | N/A |
| Safety | 2.01 to 2.26 | 2.2 to 2.4 |
| Pharmacokinetic | 3.1 to 3.3 | 3.1 to 3.3 |
| Pharmacodynamics | 4.1 to 4.2 | 4.1 to 4.4 |
| Section | Listin | Listings |
| ICH Listings | 1 to | 1 to 30 |
| Other Listings | 31 to | 31 to 33 |

### 11.8.2. Mock Example Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided in Appendix 9: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Pharmacodynamics | PD_Fn | PD_Tn | PD_Ln |

#### NOTES:

 Non-Standard displays are indicated in the 'IDSL / TST ID / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

# 11.8.3. Deliverable [Priority]

| Delivery [Priority] | Description |
|---------------------|-------------------------------------|
| SAC[1] | Final Statistical Analysis Complete |

#### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort.

# 11.8.4. Study Population Tables

| Study Pop | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] |
| Subject D | Subject Disposition | | | | |
| 1.01 | Safety | ES1 | Summary of Subject Disposition | | SAC [1] |
| 1.02 | Screened | ES6 | Summary of Screening Failures | | SAC [1] |
| 1.03 | Screened | POP_T1 | Summary of Study Analysis Populations | | SAC [1] |
| 1.04 | Safety | DV1A | Summary of Important Protocol Deviations | | SAC [1] |
| 1.05 | Safety | DV1A | Summary of Other Protocol Deviation | | SAC [1] |
| Demograp | Demographics | | | | |
| 1.06 | Safety | DM1 | Summary of Demographic Characteristics | Include BMI | SAC [1] |
| 1.07 | Safety | DM5 | Summary of Race and Racial Combinations | | SAC [1] |

# 11.8.5. Safety Tables

| Safety | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| Adver | se Events | | | | |
| 2.01 | Safety | CP_AE1p | Summary of All Adverse Events | | SAC [1] |
| 2.02 | Safety | CP_AE1p | Summary of all adverse events by maximum intensity | | SAC [1] |
| 2.03 | Safety | CP_AE1p | Summary of Drug-Related Adverse Events | | SAC [1] |
| 2.04 | Safety | CP_AE1p | Summary of all drug-related adverse events by maximum intensity | | SAC [1] |
| 2.05 | Safety | CP_AE1p | Summary of Serious Adverse Events | | SAC [1] |
| 2.06 | Safety | CP_AE1p | Summary of Adverse Events Leading to Withdrawals from Study | | SAC [1] |
| Labs | | | | | • |
| 2.07 | Safety | LB1 | Summary of Chemistry Laboratory Values | | SAC [1] |
| 2.08 | Safety | LB1 | Summary of Hematology Laboratory Values | | SAC [1] |
| 2.09 | Safety | UR3 | Summary of Urinalysis Dipstick Results | | SAC [1] |
| 2.10 | Safety | LB1 | Summary of Immonoglobulin | | SAC [1] |
| 2.11 | Safety | LB1 | Summary of Change from Baseline in Chemistry Laboratory Values | | SAC [1] |

| Safety | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 2.12 | Safety | LB1 | Summary of Change from Baseline in Hematology Laboratory Values | | SAC [1] |
| 2.13 | Safety | LB1 | Summary of Percent Change from Baseline in Immonoglobulin | Including the mean of baseline value | SAC [1] |
| 2.14 | Safety | SAFE_T1 | Worst Laboratory Toxicity Grade: Chemistry | | SAC [1] |
| 2.15 | Safety | SAFE_T1 | Worst Laboratory Toxicity Grade: Hematology | | SAC [1] |
| 2.16 | Safety | SAFE_T1 | Worst Laboratory Toxicity Grade: Urinalysis | | SAC [1] |
| 2.17 | Safety | SAFE_T1 | Worst Laboratory Toxicity Grade:<br>Immonoglobulin | | SAC [1] |
| 2.18 | Safety | SAFE_T2 | Laboratory Toxicity Grade Worsening of at Least 2 Grades from Baseline: Chemistry | | SAC [1] |
| 2.19 | Safety | SAFE_T2 | Laboratory Toxicity Grade Worsening of at Least 2 Grades from Baseline: Hematology | | SAC [1] |
| 2.20 | Safety | SAFE_T2 | Laboratory Toxicity Grade Worsening of at Least 2 Grades from Baseline: Urinalysis | | SAC [1] |
| 2.21 | Safety | SAFE_T2 | Laboratory Toxicity Grade Worsening of at<br>Least 2 Grades from Baseline:<br>Immunoglobulin | | SAC [1] |

| Safety | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| ECG | | | | | |
| 2.22 | Safety | EG2 | Summary of ECG Parameter | Use latest assessment in case of multiple assessments at any given time point | SAC [1] |
| 2.23 | Safety | EG2 | Summary of Mean Change from Baseline in ECG Values | | SAC [1] |
| 2.24 | Safety | EG1 | Summary of the Number and Percentage of Subjects Who Had Abnormal ECG Findings | Including 'Clinically Significant' and 'Not Clinically Significant' | SAC [1] |
| Vital S | igns | | | | |
| 2.25 | Safety | VS1 | Summary of Vital Signs | Including systolic blood pressure, diastolic blood pressure and pulse, respiratory Rate, temperature | SAC [1] |
| 2.26 | Safety | VS1 | Summary of Change from Baseline in Vital Signs | | SAC [1] |

# 11.8.6. Pharmacokinetic Tables

| Phari | Pharmacokinetic : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| PK C | oncentration Da | ta | | | |
| 3.1 | PK<br>Concentration | PKCT1/PK01 | Summary of Belimumab Plasma Pharmacokinetic Concentration-Time Data | | SAC [1] |
| PK P | arameter Data | | | | |
| 3.2 | PK Parameter | PKPT1/PK03 | Summary of Derived Belimumab Plasma<br>Pharmacokinetic Parameters | Including: arithmetic mean, 95% confidence interval for the arithmetic mean, standard deviation, median, minimum, maximum, between coefficient of variation, geometric mean and 95% confidence interval | SAC [1] |
| 3.3 | PK Parameter | PKPT3/PK05 | Summary of Derived Belimumab Plasma Pharmacokinetic Parameters Based on Log- Transformation | | SAC [1] |

# 11.8.7. Pharmacodynamic Tables

| Phari | Pharmacodynamic : Tables | | | | |
|---|---|---|---|---|---|
| No. Population IDSL / TST ID | | | | Deliverable [Priority] | |
| PD P | PD Parameter Data | | | | |
| 4.1 | PD | PKPT1/PK03 | Summary of B Cell Subsets | | SAC [1] |
| 4.2 | PD | PKPT1/PK03 | Summary of Percent Change from Baseline in B Cell Subsets | Including the mean of baseline value | SAC [1] |

# 11.8.8. Safety Figures

| Safet | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Responsibility<br>Deliverable [Priority] |
| Labs | | | | | |
| 2.1 | Safety | SAFE_F1 | Mean Profile of Immunoglobulin | | SAC [1] |
| 2.2 | Safety | SAFE_F1 | Median Profile of Immunoglobulin | | SAC [1] |
| 2.3 | Safety | SAFE_F2 | Mean Profile of Percent Change from Baseline in<br>Immunoglobulin | | SAC [1] |
| 2.4 | Safety | SAFE_F2 | Median Profile of Percent Change from Baseline in<br>Immunoglobulin | | SAC [1] |

Note: Use consistent colour for treatments in all figures

# 11.8.9. Pharmacokinetic Figures

| Phari | Pharmacokinetic : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Responsibility<br>Deliverable [Priority] |
| Indiv | dual Concentra | tion Plots | | | |
| 3.1 | PK<br>Concentration | PKCF1P/<br>PK16a | Individual Belimumab Plasma Concentration-Time Plot (Linear and Semi-Log) | | SAC [1] |
| Mean | Concentration | Plots | | | |
| 3.2 | PK<br>Concentration | PKCF2/ PK17 | Mean (+SD) Belimumab Plasma Concentration-Time Plot (Linear and Semi-Log) | | SAC [1] |
| Media | Median Concentration Plots | | | | |
| 3.3 | PK<br>Concentration | PKCF3/ PK18 | Median (Range) Belimumab Plasma Concentration-<br>Time Plot (Linear and Semi-Log) | | SAC [1] |

Note: Use consistent colour for treatments in all figures

# 11.8.10. Pharmacodynamic Figures

| Phari | Pharmacodynamic : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable [Priority] |
| PD P | PD Parameter Data | | | | |
| 4.1 | PD | PD_F1 | Mean Profile of B Cell Subsets | | SAC [1] |
| 4.2 | PD | PD_F1 | Median Profile of B Cell Subsets | | SAC [1] |
| 4.3 | PD | PD_F2 | Mean Profile of Percent Change from Baseline in B Cell Subsets | | SAC [1] |
| 4.4 | PD | PD_F2 | Median Profile of Percent Change from Baseline in B Cell Subsets | | SAC [1] |

# 11.8.11. ICH Listings

| ICH Lis | ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| Subjec | ct Disposition | | | | |
| 1 | Screened | ES7 | Listing of Reasons for Screening Failure | | SAC [1] |
| 2 | Safety | ES2 | Listing of Reasons for Study Withdrawal | | SAC [1] |
| 3 | Safety | DV2 | Listing of Important Protocol Deviations | | SAC [1] |
| 4 | Safety | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | SAC [1] |
| 5 | Safety | DV2 | Listing of Other Protocol Deviations | | SAC [1] |

| ICH Li | ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| Demo | graphics | | | | |
| 6 | Safety | DM2 | Listing of Demographic Characteristics | | SAC [1] |
| 7 | Safety | DM9 | Listing of Race and Racial Combinations | | SAC [1] |
| Medic | al Conditions & C | oncomitant Medica | tions | | |
| 8 | Safety | CM3 | Listing of Concomitant Medications by Generic Term | | SAC [1] |
| 9 | Safety | MH2 | Listing of Medical Conditions | | SAC [1] |
| Expos | ure | | | | |
| 10 | Safety | EX3 | Listing of Exposure | | SAC [1] |
| Adver | se Events | | | | |
| 11 | Safety | AE7 | Listings of Subject Numbers for Individual Adverse Events | | SAC [1] |
| 12 | Safety | AE2 | Relationship between System Organ Class and Verbatim Text | | SAC [1] |
| 13 | Safety | CP_AE8 | Listing of All Adverse Events | | SAC [1] |
| 14 | Safety | CP_AE8 | Listing of All Adverse Events by Maximum Intensity | | SAC [1] |
| 15 | Safety | CP_AE8 | Listing of Drug-Related Adverse Events | | SAC [1] |

| ICH Lis | ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 16 | Safety | CP_AE8 | Listing of Drug-Related Adverse Events by Maximum Intensity | | SAC [1] |
| 17 | Safety | CP_AE8a | Listing of Serious Adverse Events | The listing will be provided by fatal and non-fatal outcomes | SAC [1] |
| 18 | Safety | CP_AE8 | Listing of Adverse Events Leading to Withdrawal from Study | | SAC [1] |
| LABS | | | | | |
| 19 | Safety | SAFE_L1 | Laboratory Results: Chemistry | | SAC [1] |
| 20 | Safety | SAFE_L1 | Laboratory Results: Hematology | | SAC [1] |
| 21 | Safety | SAFE_L1 | Laboratory Results: Urinalysis | | SAC [1] |
| 22 | Safety | SAFE_L1 | Laboratory Results: Immunoglobulin | | SAC [1] |
| ECG | | | | | |
| 23 | Safety | CP_EG3 | Listing of ECG Values for All Subjects | | SAC [1] |
| 24 | Safety | CP_EG3 | Listing of All ECG Findings for Subjects with An Abnormal Finding | Including 'Clinically Significant' and 'Not<br>Clinically Significant' | SAC [1] |

| ICH Lis | ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| Vital S | Vital Signs | | | | |
| 25 | Safety | CP_VS4 | Listing of Vital Signs for All Subjects | | SAC [1] |
| Liver E | Liver Event | | | | |
| 26 | Safety | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting | | SAC [1] |
| 27 | Safety | LIVER6 | Listing of Liver Stopping Event Information for RUCAM Score | | SAC [1] |
| 28 | Safety | SAFE_L2 | Listing of Medical Conditions at Onset of Liver Event | | SAC [1] |
| 29 | Safety | LIVER7 | Listing of Liver Biopsy Details | | SAC [1] |
| 30 | Safety | LIVER8 | Listing of Liver Imaging Details | | SAC [1] |

# 11.8.12. Non-ICH Listings

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| PK | | | | | |
| 31 | PK<br>Concentration | PK08 | Listing of Individual Subject Concentration | | IA (SAC) |
| 32 | PK Parameter | PK13 | Listing of Derived Pharmacokinetic Parameters | | IA (SAC) |
| PD | | | | | |
| 33 | PD | PD_L1 | Listing of B Cell Subset | | IA (SAC) |

# 11.9. Appendix 9: Example Mock Shells for Data Displays

Data Display Specification will be made available on Request.